CLINICAL TRIAL: NCT01252888
Title: A Prospective Evaluation of Open-angle Glaucoma Subjects on Two Topical Hypotensive Medication Treated With Two Trabecular Micro-bypass Stents
Brief Title: Prospective Evaluation of Open-angle Glaucoma Subjects on Two Topical Hypotensive Medication Treated With Two iStents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCF-018
Record Dates: First submitted 2010-12-01; First posted 2010-12-03 (Estimated); Last update posted 2022-09-07 (Actual); Status verified 2017-12

CONDITIONS: Subjects With Primary Open-angle Glaucoma (POAG)
Keywords: Open angle; Glaucoma; Surgery; Glaucoma Open-Angle; Ocular Hypertension; Eye Diseases
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Two iStent devices and medication (Experimental): Implantation of two iStents through small temporal clear corneal incision
  Interventions: Device: iStents

INTERVENTIONS:
Device: iStents — Implantation of two iStents through a small temporal clear corneal incision

SUMMARY:
The purpose of this study is to assess efficacy and safety of two iStents for the reduction of intraocular pressure associated with primary open-angle glaucoma.

DETAILED DESCRIPTION:
This study evaluates the safety and efficacy of two iStents implanted in primary open-angle glaucoma subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with primary open-angle glaucoma (POAG)
* Subjects on two topical hypotensive medications

Exclusion Criteria:

* Traumatic, uveitic, neovascular, or angle closure glaucoma
* Fellow eye already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
mean diurnal IOP reduction of greater than or equal to 20% at Month 12 vs baseline | 12 months

SECONDARY OUTCOMES:
Mean diurnal IOP < 18 mmHg at month 12 | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- S.V. Malayna's Ophthalmology Centre, Yerevan, Armenia

REFERENCES:
- [Background] Ahmed II, Katz LJ, Chang DF, Donnenfeld ED, Solomon KD, Voskanyan L, Samuelson TW. Prospective evaluation of microinvasive glaucoma surgery with trabecular microbypass stents and prostaglandin in open-angle glaucoma. J Cataract Refract Surg. 2014 Aug;40(8):1295-300. doi: 10.1016/j.jcrs.2014.07.004. PMID 25088627
- [Background] Chang DF, Donnenfeld ED, Katz LJ, Voskanyan L, Ahmed II, Samuelson TW, Giamporcaro JE, Hornbeak DM, Solomon KD. Efficacy of two trabecular micro-bypass stents combined with topical travoprost in open-angle glaucoma not controlled on two preoperative medications: 3-year follow-up. Clin Ophthalmol. 2017 Mar 15;11:523-528. doi: 10.2147/OPTH.S121041. eCollection 2017. PMID 28352151